CLINICAL TRIAL: NCT03322631
Title: A Multiple-Ascending Dose Study in Japanese Patients With Type 2 Diabetes Mellitus to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY3298176
Brief Title: A Study of Tirzepatide (LY3298176) in Japanese Participants With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 16400; I8F-JE-GPGC (Other: Eli Lilly and Company)
Record Dates: First submitted 2017-10-24; First posted 2017-10-26 (Actual); Results first posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2022-06

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tirzepatide (Experimental): Participants received escalating doses of 2.5 milligrams (mg), 5 mg, 10 mg and 15 mg of tirzepatide administered into the subcutaneous (SC) tissue of the abdominal wall.
  Interventions: Drug: Tirzepatide
- Placebo (Placebo Comparator): Participants received placebo administered into the SC tissue of the abdominal wall.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tirzepatide — Administered SC.
  Other Names: LY3298176
  Arms: Tirzepatide
Drug: Placebo — Administered SC.
  Arms: Placebo

SUMMARY:
The purposes of this study are to determine:

* The safety of tirzepatide and any side effects that might be associated with it.
* How much tirzepatide gets into the bloodstream and how long it takes the body to remove it.
* How tirzepatide affects the levels of blood sugar.

This study includes eight weekly doses of tirzepatide or placebo given as subcutaneous (SC) injections just under the skin. The study will last about 16 weeks (total), including screening and follow-up. This study is for research purposes only and is not intended to treat any medical conditions.

ELIGIBILITY:
Inclusion Criteria:

* Have T2DM controlled with diet and exercise alone or are stable on a single oral antidiabetic medication (metformin or dipeptidyl peptidase [DPP]-IV inhibitors)
* Have a body mass index of 20.0 to 35.0 kilograms per square meter, inclusive

Exclusion Criteria:

* Have known allergies to tirzepatide, glucagon-like peptide (GLP)-1 analogs, or related compounds
* Have had more than 1 episode of severe hypoglycemia, as defined by the American Diabetes Association criteria, within 6 months before entry into the study or has a history of hypoglycemia unawareness or poor recognition of hypoglycemic symptoms
* Have an abnormality in the 12-lead electrocardiogram at screening that, in the opinion of the investigator, increases the risks associated with participating in the study
* Have a history or presence of pancreatitis or gastrointestinal (GI) disorder or any GI disease which impacts gastric emptying or could be aggravated by GLP-1 analogs or DPP-IV inhibitors

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2018-05-29 (Actual); Study Completion 2018-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- Japan (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Hachiōji, Tokyo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Shinjuku-Ku, Tokyo

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 2.5 mg/5 mg/10 mg Tirzepatide (Cohort 1): Participants received tirzepatide with titration regimen starting from 2.5 mg (milligrams) for Days 1 and 8 followed by 5 mg for Days 15 and 22, and 10 mg for Days 29, 36, 43, and 50 administered into the subcutaneous (SC) tissue of the abdominal wall.
- 5 mg/10 mg/15 mg Tirzepatide (Cohort 2): Participants received tirzepatide with titration regimen starting from 5 mg for Days 1 and 8 followed by 10 mg for Days 15, 22, 29, and 36, and 15 mg for Days 43 and 50 administered into the SC tissue of the abdominal wall.
- 5 mg Tirzepatide (Cohort 3): Participants received 5 mg tirzepatide administered into the SC tissue of the abdominal wall.
Period: Overall Study
Arm/Group | Placebo | 2.5 mg/5 mg/10 mg Tirzepatide (Cohort 1) | 5 mg/10 mg/15 mg Tirzepatide (Cohort 2) | 5 mg Tirzepatide (Cohort 3)
Started | 9 | 12 | 16 | 11
Received at Least 1 Dose of Study Drug | 9 | 12 | 16 | 11
Completed | 9 | 11 | 15 | 11
Not Completed | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- Placebo: Participants received placebo administered into the subcutaneous (SC) tissue of the abdominal wall.
- 2.5 mg/5 mg/10 mg Tirzepatide (Cohort 1): Participants received tirzepatide with titration regimen starting from 2.5 mg (milligrams) for Days 1 and 8 followed by 5 mg for Days 15 and 22, and 10 mg for Days 29, 36, 43, and 50 administered into the SC tissue of the abdominal wall.
- Total: Total of all reporting groups
Arm/Group | Placebo | 2.5 mg/5 mg/10 mg Tirzepatide (Cohort 1) | 5 mg/10 mg/15 mg Tirzepatide (Cohort 2) | 5 mg Tirzepatide (Cohort 3) | Total
Number analyzed (Participants) | 9 | 12 | 16 | 11 | 48
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.4 (11.6) | 56.9 (9.5) | 57.7 (8.0) | 57.5 (7.9) | 57.4 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 0 | 1
  Male | 9 | 12 | 15 | 11 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 12 | 16 | 11 | 48
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 9 | 12 | 16 | 11 | 48
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 9 | 12 | 16 | 11 | 48
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] | 22.58 (2.09) | 25.49 (2.75) | 26.10 (3.11) | 26.68 (3.29) | 25.42 (3.16)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: Safety was assessed from time of consent through end of study (up to 85 days). Data presented are the number of participants who experienced 1 or more SAEs considered by the investigator to be related to study drug. A summary of SAEs and other non-serious AEs, regardless of causality is located in the Reported Adverse Events section of this record.
Time Frame: Baseline through Day 85
Population: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 2.5 mg/5 mg/10 mg Tirzepatide (Cohort 1) | 5 mg/10 mg/15 mg Tirzepatide (Cohort 2) | 5 mg Tirzepatide (Cohort 3)
Number analyzed (Participants) | 9 | 12 | 16 | 11
Participants | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of Tirzepatide
Description: Pharmacokinetics (PK): Maximum observed drug concentration (Cmax) of Tirzepatide in plasma.
Time Frame: Predose, 8, 24, 48, 72 and 168 hours post dose for Day 1 administration, and Predose, 8, 24, 48, and 168 hours post dose for Day 50 administration
Population: All randomized participants who received at least one dose of study drug and have evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | 2.5 mg/5 mg/10 mg Tirzepatide (Cohort 1) | 5 mg/10 mg/15 mg Tirzepatide (Cohort 2) | 5 mg Tirzepatide (Cohort 3)
Number analyzed (Participants) | 11 | 12 | 11
nanograms per milliliter (ng/mL)
  Day 1 | 215 (18) | 442 (23) | 364 (20)
  Day 50 | 1520 (15) | 2270 (17) | 838 (22)

3. Secondary Outcome: PK: Area Under the Concentration Versus Time Curve (AUC) of Tirzepatide
Description: Area under the concentration versus time curve from time zero to tau (τ) of Tirzepatide (AUC[0- τ]), where tau is dosing interval of (0-168 hours).
Time Frame: as for outcome 2
Population: All randomized participants who received at least one dose of study drug and have evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms * hours per mL (ng*hr/mL)
Arm/Group | 2.5 mg/5 mg/10 mg Tirzepatide (Cohort 1) | 5 mg/10 mg/15 mg Tirzepatide (Cohort 2) | 5 mg Tirzepatide (Cohort 3)
Number analyzed (Participants) | 11 | 12 | 11
nanograms * hours per mL (ng*hr/mL)
  Day 1 | 26100 (27) | 54400 (16) | 48800 (16)
  Day 50 | 192000 (16) | 285000 (15) | 104000 (19)

4. Secondary Outcome: Pharmacodynamics (PD): Change From Baseline to 8 Weeks in Fasting Plasma Glucose
Description: Change from baseline to 8 weeks in Fasting Plasma Glucose was measured to investigate the PD effect of Tirzepatide after multiple SC doses administered to Japanese patients with T2DM
Time Frame: Baseline, Week 8
Population: All randomized participants who received at least one dose of drug and have evaluable PK data.
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)
Arm/Group | Placebo | 2.5 mg/5 mg/10 mg Tirzepatide (Cohort 1) | 5 mg/10 mg/15 mg Tirzepatide (Cohort 2) | 5 mg Tirzepatide (Cohort 3)
Number analyzed (Participants) | 9 | 11 | 15 | 11
milligram per deciliter (mg/dL) | -4.0 (23.7) | -77.5 (24.2) | -72.6 (30.9) | -51.7 (28.9)

ADVERSE EVENTS:
Time Frame: Up To 85 days
Description: All randomized participants who received at least one dose of study drug
Arm/Group | Placebo | 2.5 mg/5 mg/10 mg Tirzepatide (Cohort 1) | 5 mg/10 mg/15 mg Tirzepatide (Cohort 2) | 5 mg Tirzepatide (Cohort 3)
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/12 | 0/16 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/12 | 0/16 | 0/11
Other Adverse Events (participants affected / at risk) | 4/9 | 11/12 | 15/16 | 6/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=9) | 2.5 mg/5 mg/10 mg Tirzepatide (Cohort 1) (N=12) | 5 mg/10 mg/15 mg Tirzepatide (Cohort 2) (N=16) | 5 mg Tirzepatide (Cohort 3) (N=11)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2) | 4 (4) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (4) | 1 (1) | 0 (0) | 3 (9)
Constipation (Gastrointestinal disorders) | 1 (1) | 8 (11) | 8 (9) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 5 (7) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (4)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (3) | 2 (3) | 1 (8)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood triglycerides increased (Investigations) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 2 (4) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 6 (6) | 10 (10) | 5 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-10-15): https://cdn.clinicaltrials.gov/large-docs/31/NCT03322631/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-22): https://cdn.clinicaltrials.gov/large-docs/31/NCT03322631/SAP_001.pdf